CLINICAL TRIAL: NCT03045952
Title: Percutaneous Microwave Ablation Under Ultrasound Guidance for Primary Liver Cancer: a Multicenter Analysis
Brief Title: Percutaneous Microwave Ablation Under Ultrasound Guidance for Liver Cancer: a Multicenter Analysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Professor, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 66939530lp
Record Dates: First submitted 2016-12-26; First posted 2017-02-08 (Estimated); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Liver Neoplasms
Keywords: Multicenter study; microwave
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- microwave ablation (Experimental): Antenna in the microwave ablation device was percutaneously inserted into the tumor and placed at designated place under US guidance. For tumors less than 1.5 cm, one antenna was inserted and for tumors measuring 1.5 cm or greater, two antennae were inserted in parallel with an inter-antenna distance of 1.0-2.5 cm, which were used simultaneously during MWA to obtain larger ablation zone. A 20G thermocouple was inserted about 0.5-1 cm away from the tumor for real-time temperature monitoring during MWA. MW emission didn't stop until the heat-generated hyperechoic water vapor completely encompassed the entire tumor and the measured temperature reached 60°C or remained above 54°C for at least three minutes.
  Interventions: Procedure: microwave ablation device

INTERVENTIONS:
Procedure: microwave ablation device — Microwave ablation is a technique that uses thermal therapy to induce complete necrosis of tumor in situ by using microwave ablation device.

SUMMARY:
Ultrasound-guided percutaneous MWA of liver cancer is a relatively new technique with favorable long-term outcomes.Butthe results are mainly from single center reports.A larger scale data need to be analyzed to evaluate the technique. This study is designed to investigated the efficacy of cooled-tip microwave ablation (MWA) for primary liver cancer (PLC) and analyzed the prognostic factors on a multicenter database.Between January 2013 and December 2018, all the PLC patients underwent ultrasound-guided percutaneous cooled-tip MWA as a primary treatment will be enrolled from at least ten Chinese institutions with different levels of MWA experience. All the patients will be closely followed up until June 2019. Clinicopathologic data, recurrence and survival estimates, complications and prognosis-relative factors will be measured.

ELIGIBILITY:
Inclusion Criteria:

* absence of ascites or the depth of ascites on US detection less than 4 cm;
* a normal serum total bilirubin level or less than 60 µmol/L;
* a normal albumin level or not less than 30 g/L;
* for radical treatment, single lesion of 8 cm or smaller, three or fewer multiple lesions with a maximum diameter of 4 cm or less, absence of portal vein cancerous thrombus or extrahepatic metastases;
* for palliative treatment, those with large or multiple lesions, suffering multiple metastases and unsuitable for other modalities can be considered to undergo the MWA on the condition of good hepatic function and blood coagulation function to tolerate the procedure.

Exclusion Criteria:

Contraindications include patients who have

1. clinical evident liver failure, such as massive ascites or hepatic encephalopathy or with a trance-like state;
2. severe blood coagulation dysfunction (prothrombin time of more than 30 seconds, prothrombin activity less than 40%, and platelet count less than 30 cells×109/L);
3. high intrahepatic tumor burden (tumor volume >70% of the target liver volume or multiple tumor nodules) or high extrahepatic tumor burden;
4. acute or active inflammatory and infectious lesions at any organ;
5. acute or severe chronic renal failure, pulmonary insufficiency or heart dysfunction;
6. relative contraindication concerns medical risk for the tumor proximity to diaphragm, gastrointestinal tract, gallbladder, pancreas, hepatic hilum and major bile duct or vessels, which may require adjunctive techniques to prevent off-target heating of adjacent structures during the ablation procedure.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1908 (Actual)
Dates: Start 2013-01; Primary Completion 2019-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
overall survival | 5 years

SECONDARY OUTCOMES:
intrahepatic metastasis | 5 years
extrahepatic metastasis | 5 years
local tumor progress | 5 years
complication | 1 month
  number of participants with side effect and major complication
disease free survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, Dr., Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cai Q, Pang C, Wang Z, Li J, Dai Y, Fan FY, Wang ZQ, Hu X, Li L, Chen XW, Ji R, Mei Q, Zhang C, Liang P, Yu X, Liu FY, Cheng Z, Yu J. Relationship between postablation fever and prognosis in initial hepatocellular carcinoma: a 15-year multicenter, retrospective cohort study. Int J Surg. 2025 Jan 1;111(1):962-971. doi: 10.1097/JS9.0000000000002066. PMID 39291970